CLINICAL TRIAL: NCT02769078
Title: Replication Of An Early Evaluation Of 30-Day Readmissions Among Nonvalvular Atrial Fibrillation Patients Treated With Dabigatran, Rivaroxaban, Apixaban, or Warfarin In The U.S
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-425
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Atrial Fibrillation
Keywords: Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Rivaroxaban; apixaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients who received dabigatran: Patients who received dabigatran
  Interventions: Drug: dabigatran
- Patients who received rivaroxaban: Patients who received rivaroxaban
  Interventions: Drug: rivaroxaban
- Patients who received apixaban: Patients who received apixaban
  Interventions: Drug: apixaban
- Patients who received warfarin: Patients who received warfarin
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: dabigatran
  Groups: Patients who received dabigatran
Drug: rivaroxaban
  Groups: Patients who received rivaroxaban
Drug: apixaban
  Groups: Patients who received apixaban
Drug: warfarin
  Groups: Patients who received warfarin

SUMMARY:
The overall objective of this proposal is to execute a real-world database analysis to evaluate hospital readmissions among hospitalized nonvalvular atrial fibrillation (NVAF) patients in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary or secondary diagnosis of AF identified by International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) codes from the Cerner Health Facts hospital database between January 1, 2012 and August 31, 2014
* Age 18 years or older as of initial hospitalization with AF diagnosis

Exclusion Criteria:

* Have any primary or secondary diagnosis code or procedure code for valvular disease during the study period. This exclusion criterion is consistent with that used in other previous BMS Health Economics and Outcomes Research (HEOR) studies and is used to ensure that the study populations are NVAF patients
* Received multiple types of NOACs during the index hospitalization. Preliminary analysis showed that very few patients receive multiple types of NOACs during the same hospitalization. This exclusion criterion will allow to cleanly group patients into the different New oral anticoagulant (NOAC) usage groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received any of the NOACs, dabigatran, rivaroxaban, apixaban, or warfarin during any time of the hospitalization (from admission to discharge)
Sampling Method: Non-Probability Sample
Enrollment: 14201 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of NVAF patients with bleeding-related hospital readmissions from inpatient hospitalization records collected from the Cerner Health Facts hospital database | January 1, 2012 to August 31, 2014
  Proportion of NVAF patients with bleeding-related hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban, or warfarin in the inpatient setting.

SECONDARY OUTCOMES:
Cost associated with bleeding-related hospital readmissions from inpatient hospitalization records collected from the Cerner Health Facts hospital database | January 1, 2012 to August 31, 2014
  Cost associated with bleeding-related hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban, or warfarin in the inpatient setting
Proportion of NVAF patients with all cause hospital readmissions and the associated costs from inpatient hospitalization records collected from the Cerner Health Facts hospital database | January 1, 2012 to August 31, 2014
  Proportion of NVAF patients with all cause hospital readmissions and the associated costs that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban, or warfarin in the inpatient setting.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx